CLINICAL TRIAL: NCT05788211
Title: Predicted Long Term Renal Outcome After Medical or Postcardiotomy Refractory Cardiogenic Shock Requiring Renal Replacement Therapy Concomitant With Venoarterial Extracorporeal Membrane Oxygenation
Brief Title: REnal reCOVery After ECMO for Cardiogenic Shock (RECOVECMO)
Acronym: RECOVECMO
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Principal Investigator, Alexandre OUATTARA, Head of department of Cardiovascular Anesthesia and Critical care, University Hospital, Bordeaux
Other Study IDs: SAR CV 1
Record Dates: First submitted 2023-02-24; First posted 2023-03-28 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Cardiogenic Shock; Renal Replacement Therapy; Venoarterial Extracorporeal Membrane Oxygenation
Keywords: Cardiogenic shock; Renal replacement therapy; venoarterial extracorporeal membrane oxygenation; extra corporeal life support; major adverse kidney events; acute kidney injury; end-stage renal disease; serum creatinine
MeSH Terms: conditions — Shock, Cardiogenic; Acute Kidney Injury; Kidney Failure, Chronic | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- REFRACTORY CARDIOGENIC SHOCK: All patients with medical or postcardiotomy refractory cardiogenic shock requiring renal replacement therapy concomitant with venoarterial extracorporeal membrane oxygenation.
  Interventions: Other: standard of care

INTERVENTIONS:
Other: standard of care — retrospective study: standard of care

SUMMARY:
This retrospective study assesses long term renal outcome in patients having suffered medical or post cardiotomy refractory cardiogenic shock requiring renal replacement therapy (RRT) concomitant with veno-arterial extracorporeal membrane oxygenation (VA-ECMO).

The authors seek to establish for accurate definition of renal recovery status predicting poor long-term renal outcomes.

DETAILED DESCRIPTION:
Cardiogenic shock, defined as cardiac pump failure, is caused by many etiologies such as myocardial infarction, infectious diseases or post-cardiotomy. Mortality remains high and may reach 80% depending on etiologies and series ( 60% 30 days - mortality after post-cardiotomy cardiogenic shock). Extra Corporeal Life Support (ECLS) became a corner stone of refractory cardiogenic shock.

This low cardiac output syndrome leeds to associated organs failure whose renal function is the first being impaired. Severity partly depends on hemodynamic instability duration and intensity. Sixty percent of patients under ECLS develop acute kidney injury (AKI) and two third of them will need renal replacement therapy (RRT), representing 40 percent of the ECLS population. In addition, RRT introduction is associated with higher mortality.

In the surviving patients, there is a growing interest on long term renal outcomes. Few retrospective studies already indicate a higher 1- and 2-years incidence of major adverse kidney events (MAKE: overall mortality or dialysis dependance or doubling serum creatinine) in case of association of RRT and ECLS. Also, 90 days renal recovery status may be correlated with 2.9 higher risk of MAKE at 3 years.

Nowadays, preventing those long term renal adverse events should be considered as a priority during intensive care unit stay. Optimizing renal recovery appears to be the leading strategy in clinical practice.

There is a lack of standardization in defining renal recovery leading to incomparability of studies. To investigators knowledge, there is no validated definition of renal recovery in patients undergoing combined veno-arterial mode of extracorporeal oxygenation membrane (VA mode of ECMO) and renal replacement therapy.

The RECOVECMO study proposes to determinate the sensitivity and specificity of two definitions of renal recovery (serum creatinine level below 1.5 fold serum creatinine basal level or serum creatinine level below 1.25 fold serum creatinine basal level) in predicting 2 years incidence of MAKE in patients undergoing renal replacement therapy while receiving VA mode of ECMO.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Medical or post cardiotomy refractory cardiogenic shock
* Patients requiring concomitant renal replacement therapy (RRT) and venoarterial extracorporeal membrane oxygenation (VA-ECMO)

Exclusion Criteria:

* Congenital heart diseases
* Severe pre operative chronic kidney disease (eGFR < 30ml/min/1,73m2)
* Death within the first 7 days of ECMO
* Patient receiving non-concomitant ECMO and RRT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients having suffered of medical or post cardiotomy refractory cardiogenic shock requiring renal replacement therapy concomitant with venoarterial extracorporeal membrane oxygenation, and meeting the protocol criteria between 2012, january the first and 2020, june the first.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Complete renal recovery status according first definition | 90 days from AKI (acute Kidney Injury) start
  decrease in serum creatinine level below 1.5 fold its basal value
Complete renal recovery status according second definition | 90 days from AKI start
  decrease in serum creatinine level below 1.25 fold its basal value
Long term renal outcome | 2 years from AKI start
  proportion of patient meeting a composite criterion (overall mortality or dialysis dependency or doubling of basal serum creatinine)

SECONDARY OUTCOMES:
MAKE incidence | 7 days , 90 days, 1 year , 2 years from AKI start
  Major Adverse Kidney Events incidence: death or dialysis dependency or serum creatinine value ≥ 200 % of the baseline serum creatinine.
MAKE incidence | hospital discharge, an average of 60 days from AKI start
  Major Adverse Kidney Events incidence: death or dialysis dependency or serum creatinine value ≥ 200 % of the baseline serum creatinine.
Renal recovery status | 7 days , 90 days, 1 year , 2 years from AKI start
  Renal recovery status through serum creatinine measure
Renal recovery status | hospital discharge, an average of 60 days from AKI start
  Renal recovery status through serum creatinine measure
vital status | 1 year, 2 years from AKI start
  Mortality from AKI start
renal replacement therapy status | 1 year, 2 years from AKI start
  number of patients requiring renal replacement therapy assessed thanks to medical records
Determination of risk factors (baseline characteristics, clinical features, medications and nephrotoxic use, ECMO parameters, RRT parameters) associated with incomplete renal recovery status | up to 90 days from AKI start
  Report data (baseline characteristics, clinical features, medications and nephrotoxic use, ECMO parameters, RRT parameters) present at inclusion or appearing during the follow-up of patients who have not completely recovered their renal function 90 days after the start of AKI
Determination of risk factors (baseline characteristics, clinical features, medications and nephrotoxic use, ECMO parameters, RRT parameters, 90 days renal recovery status) associated with MAKE | up to 2 years from AKI start
  Report data present at inclusion or appearing during the follow-up of patients (baseline characteristics, clinical features, medications and nephrotoxic use, ECMO parameters, RRT parameters, 90 days renal recovery status) associated with MAKE, up to 2 years after the start of AKI

CONTACTS AND LOCATIONS:
Locations (1):
- Bordeaux University Hospital, Pessac, France

REFERENCES:
- [Background] Bellomo R, Ronco C, Kellum JA, Mehta RL, Palevsky P; Acute Dialysis Quality Initiative workgroup. Acute renal failure - definition, outcome measures, animal models, fluid therapy and information technology needs: the Second International Consensus Conference of the Acute Dialysis Quality Initiative (ADQI) Group. Crit Care. 2004 Aug;8(4):R204-12. doi: 10.1186/cc2872. Epub 2004 May 24. PMID 15312219
- [Background] Pannu N, James M, Hemmelgarn B, Klarenbach S; Alberta Kidney Disease Network. Association between AKI, recovery of renal function, and long-term outcomes after hospital discharge. Clin J Am Soc Nephrol. 2013 Feb;8(2):194-202. doi: 10.2215/CJN.06480612. Epub 2012 Nov 2. PMID 23124779